CLINICAL TRIAL: NCT05410704
Title: Effects of Pelvic Floor Muscle Training and Diaphragmatic Breathing Exercise Via Telerehabilitation on Body Posture and Quality of Life Outcomes
Brief Title: Effects of Pelvic Floor Muscle Training and Diaphragmatic Breathing Exercise on Body Posture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: postureandlife
Record Dates: First submitted 2022-05-28; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Telerehabilitation; Body Posture; Pelvic Floor Muscle Training; Diaphragmatic Breathing; Quality of Life
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Pelvic floor muscle exercises and diaphragmatic breathing exercises will be performed 3 times a week for 12 weeks. New York Posture Rating Scale and SF-36 will be applied before and after the study. International Physical Activity Questionnaire and Pelvic Floor Impact Questionnaire will be applied before the study.
  Interventions: Other: exercises
- Control Group (No Intervention): No intervention. New York Posture Rating Scale and SF-36 will be applied before and after the study. International Physical Activity Questionnaire and Pelvic Floor Impact Questionnaire will be applied before the study.

INTERVENTIONS:
Other: exercises — Pelvic floor muscle exercises and diaphragmatic breathing exercise
  Arms: Study Group

SUMMARY:
This study; It will be done in order to show evidence of the effects of pelvic floor muscle training and diaphragmatic breathing exercise via telerehabilitation on body posture and quality of life in healthy individuals. International Physical Activity Quastionnaire Short Form (IPAQ), Pelvic Floor Impact Quastionnaire Short Form (PFIQ-7), 36-Item Short Form Survey(SF-36) and New York Posture Rating Chart will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18-25
* Being a woman over the age of 18

Exclusion Criteria:

* obstructive or restrictive lung disease
* diagnosed with urinary incontinence or pelvic organ prolapse
* pelvic pain
* history of pelvic surgery
* Any history of spinal, thoracic or abdominal surgery
* To smoke
* cardiac, neurological and rheumatological disease
* Congenital deformity or previous history of surgery in the spine and thorax
* endocrine and metabolic disease
* psychiatric disorders
* cardiological disorders
* malignancy
* Doing regular physical activity or sports for the last 3 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Quality of Life | baseline
  36-Item Short Form Survey (SF-36). On the scale, higher scores mean a better outcome. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight.
Assessment of Body Posture | baseline
  New York Posture Rating Chart. On the scale, each body segment was scored 5 (correct posture), 3 (slight deviation), or 1 (pronounced deviation). The scores of the body alignment segments are summed, allowing a range of overall score between 13 and 65. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Assessment of Physical Activity Level | baseline
  International Physical Activity Questionnaire-short form (IPAQ-SF) The questionnaire records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting.
Assessment of Pelvic Floor Muscle Function | baseline
  Pelvic Floor Impact Questionnaire (PFIQ). The PFIQ 7 has 7 questions and each question has 3 separate responses. The response to each item of satisfaction, impact and worry was rated from 3 (quite a bit) to 0 (not at all) for the PFIQ-7. The mean value for all the answered items within the corresponding scale (possible value 0-3) was estimated, then multiplied by (100/3) to obtain the scale score, range 0-100. We added the scores from the 3 scales together to obtain the PFIQ 7 summary score (range 0-300).For the scale, a higher score indicates worse health status.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem VURAL, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Tülay Ülkü SEVİM, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No